CLINICAL TRIAL: NCT00622466
Title: Phase II Trial of Sorafenib and Paclitaxel for Measurable Metastatic HER2-Negative Breast Cancer
Brief Title: Sorafenib and Paclitaxel in Treating Patients With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study sponsor requested that the study be permanently closed by letter.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Barbara Haley, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 082010-161; ONYX-SCCC-112007-035; CDR0000587470 (Registry Identifier: PDQ (Physician Data Query)); NCI-2011-02791 (Registry Identifier: CTRP (Clinical Trials Reporting System))
Record Dates: First submitted 2008-02-22; First posted 2008-02-25 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer; HER2-negative breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Paclitaxel; Albumin-Bound Paclitaxel; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorfenib + Paclitaxel (Experimental): Oral sorafenib tosylate twice daily on days 1-28 and paclitaxel IV over 1 hour on days 1, 8, and 15
  Interventions: Drug: paclitaxel; Drug: sorafenib tosylate

INTERVENTIONS:
Drug: paclitaxel — The chemotherapy drug called paclitaxel (Taxol) treats breast cancer, lung cancer, ovarian cancer and Kaposis sarcoma
  Other Names: Taxol, Abraxane, Onxol
Drug: sorafenib tosylate — Sorafenib is a type of targeted therapy known as a kinase inhibitor used to treat advanced renal cell carcinoma and unresectable hepatocellular carcinoma
  Other Names: Nexavar

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving sorafenib together with paclitaxel may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving sorafenib together with paclitaxel and to how well it works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the efficacy of sorafenib tosylate and paclitaxel by measuring tumor response, as defined by RECIST criteria, in patients with metastatic, HER2-negative breast cancer.

Secondary

* To evaluate time to disease progression in patients treated with this regimen.
* To evaluate six-month progression-free survival of patients treated with this regimen.
* To evaluate time to treatment failure in patients treated with this regimen.
* To evaluate clinical benefit rate (tumor response and stable disease) at 24 weeks in patients treated with this regimen.
* To evaluate duration of response in patients treated with this regimen.
* To evaluate the tolerability of this regimen in these patients.
* To examine the relationship of gene expression and tissue/serum protein markers, where available, related to response to therapy focusing on growth factor receptor pathways.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib tosylate twice daily on days 1-28 and paclitaxel IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 4 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Histologically* confirmed breast cancer

  * Stage IV (metastatic) disease

    * Radiographic evidence of metastases NOTE: *Histological confirmation of the actual metastasis is not required.
* Measurable disease by RECIST criteria defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques (i.e., physical examination, CT scan, MRI, or x-ray) or ≥ 10 mm by spiral CT scan

  * No prior radiotherapy unless growth has been documented following radiotherapy
* Primary tumor or metastatic tumor HER2-negative, defined as the following:

  * Immunohistochemistry of 0 or 1+ OR the equivalent, if an automated quantitative assay is used
  * HER2 fluorescent in situ hybridization (FISH) assay negative as defined by a HER2:chromosome 17 centromeric probe ratio < 1.8 (or < 2.2 if immunohistochemistry is less than 3+ or equivalent) OR equivalent values for negative FISH assays that do not normalize to chromosome 17
* Hormone-receptor positive (estrogen receptor-[ER] or progesterone receptor [PgR]-positive) disease or hormone receptor-negative (ER- or PgR-negative) disease
* Tumor block from initial breast cancer primary or a biopsy of a metastatic site must be available for correlative studies
* Brain metastases allowed provided the patient is stable after completion of treatment (i.e., surgery and/or radiotherapy), asymptomatic, and off steroids with 2 consecutive stable brain scans at least 4 weeks after radiotherapy

Exclusion criteria:

* Bone-only or other nonmeasurable-only disease
* Newly diagnosed brain metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-1
* Life expectancy > 6 months
* Menopausal status not specified
* WBC ≥ 3,000/mcL
* Absolute neutrophil count ≥ 1,500/mcL
* Platelets ≥ 100,000/mcL
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT transaminases ≤ 2.5 times ULN (< 5 times ULN if liver involvement)
* Creatinine < 1.5 times ULN OR creatinine clearance > 60 mL/min
* INR < 1.5 OR PT/PTT normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to and during (women and men) and for at least 3 months after (men) study therapy
* Able to swallow and absorb oral medications

Exclusion criteria:

* Active or uncontrolled medical illness (e.g., active infection > CTCAE grade 2), including any of the following:

  * HIV or chronic hepatitis B or C
  * Uncontrolled diabetes
  * NYHA class II-IV uncompensated congestive heart failure
  * Unstable angina (anginal symptoms at rest)
  * New onset angina (i.e., began within the past 3 months)
  * Coronary artery disease
* Myocardial infarction within the past 6 months
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis or coagulopathy
* Pulmonary hemorrhage/bleeding event > CTCAE grade 2 within 4 weeks of first dose of study drug
* Any other hemorrhage/bleeding event > CTCAE grade 3 within 4 weeks of first study drug
* Thrombotic or embolic events (i.e., cerebrovascular accident), including transient ischemic attacks within the past 6 months
* Hypertension that cannot be controlled with medication to ≤ 150/90 mm Hg
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to sorafenib tosylate
* Prior invasive cancer other than breast cancer except nonmelanoma skin cancer
* Chronic nonhealing wound or ulcer

PRIOR CONCURRENT THERAPY:

* No more than 1 prior chemotherapy regimen for metastatic breast cancer (MBC)
* At least 3 weeks since prior hormonal therapy for MBC or adjuvant or neoadjuvant chemotherapy

  * More than 1 year since adjuvant paclitaxel
* At least 4 weeks since major thoracic, abdominal, or pelvic surgery and recovered
* At least 3 weeks since prior and no concurrent investigational drugs
* Concurrent bisphosphonates allowed
* Concurrent anticoagulation agents (i.e., warfarin or heparin) allowed
* No anticipated need for or concurrent radiotherapy
* No concurrent Hypericum perforatum (St. John wort) or rifampin (rifampicin)
* No other concurrent anti-neoplastic drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04-23 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B. Haley, MD, Principal Investigator — Simmons Cancer Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sorfenib + Paclitaxel
Started | 20
Completed | 16
Not Completed | 4
Not completed — Death | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression
Description: Progression-free survival was defined as the time of treatment to the earliest date of documentation of disease progression or death due to any cause. In the case of a participant started treatment. Tenth month of progression-free rate of sorafenib and paclitaxel will be compared agains the null progression free rate of 32% using normal approximation test.
Time Frame: Time from first treatment to disease progression or death (up to 36 months)
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 16
months | 6.6 [4.5 to 7.5]

2. Secondary Outcome: Tumor Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT and MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions. The confirmed response rate was estimated by the number of confirmed responses divided by the total number of participants randomized.
Time Frame: Up to 36 months
Measure: Number; unit: % of participants
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 16
% of participants | 18.75

3. Secondary Outcome: Six-month Progression-free Survival
Description: The proportion of patients with progression-free survival at 6 months. Progression-free is measured from Day-1 of study drug administration to disease progression as defined by Response Evaluation Criteria in Sole Tumors (RECIST) v1.1, or death on study. Progression is defined in RECIST v1.1 as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new leasions.
Time Frame: 6 months
Population: This data were not collected.
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 0

4. Secondary Outcome: Time to Treatment Failure
Description: Number of patients experiencing treatment failure.
Time Frame: Up to 36 months
Population: This data were not collected.
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 0

5. Secondary Outcome: Clinical Benefit Rate (Tumor Response and Stable Disease) at 24 Weeks
Description: Number of patients with either complete response (CR) or partial response (PR) as defined in Response Evaluation Criteria in Solid Tumors (for patients with measurable disease). Complete Response: Disappearance of all target lesions, disappearance of all non-target lesions for at least 4 weeks. Partial Response: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameters.
Time Frame: 24 weeks
Population: This data were not collected.
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 0

6. Secondary Outcome: Duration of Response
Description: Number weeks until disease progression measured from Day-1 of study drug administration to disease progression.
Time Frame: Up to 36 months
Population: This data were not collected.
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 0

7. Secondary Outcome: Tolerability of Sorafenib/Paclitaxel Regimen
Description: Number of patients without experiencing treatment-related adverse events.
Time Frame: Up to 36 months
Population: This data were not collected.
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 0

8. Secondary Outcome: Determine the Relationship of Gene Expression and Tissue/Serum Protein Markers, Where Available, Related to Response to Therapy Focusing on Growth Factor Receptor Pathways.
Description: Median values taken for all assays at baseline and relationship to response vs. no response will be made to identify predictive markers using methods to detect differential expression between two groups samples, including variants of the two-sample t-test, analysis of variance, F-test, and the Wilcoxon rank-sum test.
Time Frame: Up to 36 months
Population: This data were not collected.
Arm/Group | Sorfenib + Paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Weekly until end of study, as average of up to 36 months
Arm/Group | Sorfenib + Paclitaxel
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 11/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorfenib + Paclitaxel (N=16)
Gangrene wound (Infections and infestations) | 1 (1) — Grade 3 Gangrene wound
Diarrhea (Gastrointestinal disorders) | 1 — Grade 3 Diarrhea
Fatigue (General disorders) | 2 (2) — Grade 3 Fatigue
Hand-foot (Infections and infestations) | 5 (5) — Grade 3 Hand-foot
Hypertension (Cardiac disorders) | 1 (1) — Grade 3 Hypertension
Nausea/vomiting (Gastrointestinal disorders) | 1 (1) — Grade 3 Nausea/vomiting
Asymptomatic pulmonary emboli (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 4 Asymptomatic pulmonary emboli

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No